CLINICAL TRIAL: NCT05768711
Title: Phase II Study With Safety run-in of Azacitidine (AZA) Combined With Venetoclax (VEN) in Patients With Higher-risk Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Azacitidine Combined With Venetoclax in Patients With Higher-risk Chronic Myelomonocytic Leukemia (AVENHIR)
Acronym: AVENHIR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVENHIR; 2024-514878-53-00 (EU CTIS Number); 2021-002007-35 (EudraCT Number)
Record Dates: First submitted 2023-02-23; First posted 2023-03-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CMML; Azacitidine; Venetoclax
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacidine+Venetoclax (Experimental): Azacitidine will be administered subcutaneously at the standard dose of 75 mg/m²/d either on days 1-7 or using a 5-2-2 schedule of the 28 day-cycles.
  Patiens will be exposed to Venetoclax during the first 7 or 14 days of the 28 day-cycles (number of days of Venetoclax determined during the safety run-in phase).
  At cycle 1, Venetoclax will be given orally with 3-day ramp-up, at 100 mg on day 1, 200 mg on day 2 and 400 mg on days 3 to 7 or 14 of the cycle.
  At all subsequent cycles, Venetoclax will be given orally at 400 mg on days 1 to 7 or 14 of the cycle.
  Treatment duration will be 24 months.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Combination of Azacitidine and Venetoclax
  Other Names: ABT-199

SUMMARY:
Open-label phase II, single arm, multicenter study with safety run-in to evaluate the efficacy and safety of Azacitidine combined with Venetoclax in patients with higher-risk chronic myelomonocytic leukemia

DETAILED DESCRIPTION:
AVENHIR trial is an open-label phase II, single arm, multicenter study with safety run-in to evaluate the efficacy and safety of the combination of Azacitidine and Venetoclax in, hypomethylating agent-naïve, higher-risk chronic myelomonocytic leukemia patients

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older.
2. CMML diagnosis according to ICC 2022 criteria.
3. Intermediate-2 or high risk according to the molecular CMML Prognostic Scoring System (CPSS-mol) at study entry. In patients treated with HY at screening, the white blood count (WBC) prior to introduction of HY will be used to compute CPSS-mol. In patients with failed or missing cytogenetics or genetics at screening, cytogenetics and genetics at CMML diagnosis will be used to compute CPSS-mol.
4. No prior treatment with hypomethylaing agents, including Azacitidine, decitabine, SGI-110, AST7227 or CC-486 for CMML or any antecedent condition, including antecedent MDS or auto-immune disease. Prior treatment with Erythropoiesis Stimulating Agents (ESA) is allowed with a > 15 days washout from ESAs. Prior treatment with hydroxyurea (HY) is acceptable. No washout is necessary for those patients but pre-HY WBC will be taken in consideration for CPSS-mol computation.
5. Performance status 0-2 on the Eastern Cooperative Oncology Group (ECOG) Scale.
6. Adequate organ function including the following:

   * total bilirubin < 2 times upper limit of normal (ULN) (except moderate unconjugated hyperbilirubinemia due to intra medullary hemolysis or due to Gilbert syndrome),
   * alanine transaminase (ALT) and aspartate transaminase (AST) < 3 times ULN,
   * Creatinine clearance > 30 mL/min as estimated by the CKD-EPI equation.
7. Signed Informed Consent Form (ICF).
8. Negative pregnancy and adequate contraception (including in male patients) if relevant.

   A FCBP (female of childbearing potential) for this study is defined as a sexually mature woman who: (1) has not undergone a hysterectomy or bilateral oophorectomy; or (2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).

   A FCBP participating in the study must:
   * Have had 2 negative pregnancy tests as verified by the investigator prior to starting investigational medicinal product (IMP) (unless the screening pregnancy test was done within 72 hours of Cycle 1 Day 1). She must have had agreed to ongoing pregnancy testing during the course of the study and after end of treatment.
   * If sexually active, agree to use, and be able to comply with, highly effective contraception** without interruption, 5 weeks prior to starting IMP, during treatment with IMP (including dose interruptions), and for 3 months after the last dose of IMP.

     * Highly effective contraception is defined in this protocol as the following (information also appears in the ICF): Hormonal contraception (eg, birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation (tying your tubes), or a partner with a vasectomy.

   Male subjects must have agreed to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (eg, polyurethane), during sexual contact with a pregnant female or a FCBP while participating in the study, during dose interruptions, and for at least 3 months after the last dose of IMP, even if he had undergone a successful vasectomy.
9. Affiliation to a health insurance system.

Exclusion Criteria:

1. Myeloproliferative / myelodysplastic syndrome other than CMML.
2. Bone marrow or peripheral blood blasts (including promonocytes) ≥ 20%. If both local and central review are available and discrepant, the central review will be used.
3. CMML with t(5;12) or PDGFRbeta rearrangement that may be treated with imatinib.
4. Unavailable CPSS-mol at inclusion (WBC prior to HY used to compute CPSS-mol at inclusion in HY-exposed patients) or with a CPSS-mol low or intermediate-1 at study entry.
5. Pregnant or breastfeeding.
6. Serious concomitant systemic disorder, including auto-immune or auto-inflammatory disease requiring > 20 mg/d prednisone equivalent, active bacterial, fungal or viral infection that in the opinion of the investigator, would compromise the safety of the patient and/or his/her ability to complete the study.
7. Medical condition requiring therapies with CYP3A strong or moderate inducing or inhibiting activity at screening. All strong or moderate CYP3A inducers should be discontinued 7 days prior to the first dose of study drug. All strong or moderate CYP3A inhibitors should be discontinued 3 days prior to the first dose of study drug. A sample list of CYP3A4 inhibitors and inducers is provided in Appendix F.
8. Prior malignancy (except in situ cervix carcinoma, limited basal cell carcinoma, asymptomatic prostatic cancer not requiring treatment, or other tumors if not active during the last 2 years).
9. Known positive test for human immunodeficiency virus (HIV). Note that HIV testing is not required at Screening.
10. Malabsorption syndrome or other condition that precludes an enteral route of administration.
11. Previous therapy with a hypomethylating agent including azacitidine, decitabine, SGI-110, AST7227 or CC-486 for CMML or any antecedent condition, including antecedent MDS or auto-immune disease.
12. Previous therapy with a BH3 mimetic.
13. Antecedent allogeneic stem cell transplantation (HSCT) for CMML or an antecedent of hematological malignancy. Those never transplanted but eligible for HSCT are eligible for the trial.
14. Subjects referred to in Articles L1121-5 to L1121-8-1 and L1122-1-2 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Safety run-in | after 2 cycles of treatment of the safety run-in phase patients (each cycle is 28 days)
  Determination of dose-limiting toxicities within the first two cycles of treatment
Overall response rate | after 3 and 6 cycles of treatment of the phase II patients (each cycle is 28 days)
  Overall response encompasses complete remission, partial remission, marrow response and clinical benefit according to protocol-defined criteria modified from MDS/MPN IWG criteria after 3 and 6 cycles of treatment

SECONDARY OUTCOMES:
Complete remission rate | after 3 and 6 cycles of treatment (each cycle is 28 days)
  Complete remission according to protocol-defined criteria modified from MDS/MPN IWG criteria after 3 and 6 cycles of treatment
Overall response rate at best response | through study completion, an average of 5 years
  Overall response (complete remission, partial remission, marrow response, clinical benefit) according to protocol-defined criteria modified from MDS/MPN IWG criteria at best response
Overall response rate after 3 and 6 cycles of treatment | after 3 and 6 cycles of treatment (each cycle is 28 days)
  Overall response (complete remission, partial remission, marrow response, clinical benefit) according to the DACOTA trial response criteria after 3 and 6 cycles of treatment
Duration of response | through study completion, an average of 5 years
  Duration of response defined as the time interval between the first date of achievement of any response according to MDS/MPN IWG criteria to progressive disease
Identification and grading of adverse events | through study completion, an average of 5 years
  Safety profile, both hematological and non-hematological of treatment (Venetoclax combined with Azacitidine) including identification and grading of adverse events based on NCI CTCAE version 5.0
Overall survival | through study completion, an average of 5 years
  Overall survival defined as the time from inclusion until death or end of follow-up
Acute Myeloid Leukemia (AML)-free survival | through study completion, an average of 5 years
  AML-free survival defined as the time from inclusion to transformation to AML according to WHO 2016 criteria, death or end of follow-up, whichever occurs first
Progression-free survival | through study completion, an average of 5 years
  Progression-free survival defined as the time from inclusion to progressive disease according to MDS/MPN IWG criteria, transformation to AML, death or end of follow-up, whichever occurs first
Event-free survival | through study completion, an average of 5 years
  Event-free survival defined as the time from inclusion to failure to achieve any response according to MDS/MPN IWG criteria at the 6-cycle evaluation, occurence of progressive disease according to MDS/MPN IWG criteria, transformaion to AML, or death, whichever occurs first
Cumulative incidence of AML and cumulative risk of death without AML | through study completion, an average of 5 years
  Cumulative incidence of AML and cumulative risk of death without AML, considering death and transformation to AML as competing risk
Cumulative incidence of progressive disease or transformation to AML and cumulative risk of death without progression or AML | through study completion, an average of 5 years
  Cumulative incidence of progressive disease or transformation to AML and cumulative risk of death without progression or AML
Rate of Hematopoietic Stem Cell Transplantation (HSCT) | through study completion, an average of 5 years
  Rate of Hematopoietic Stem Cell Transplantation (HSCT) and post-HSCT ovrall survival and AML-free survival
Survival censoring at Hematopoietic Stem Cell Transplantation (HSCT) | through study completion, an average of 5 years
  Overall survival, AML-free survival and progressive-free survival censoring at Hematopoietic Stem Cell Transplantation (HSCT)
Subsequent therapy | through study completion, an average of 5 years
  Rate and description of subsequent therapy
Survival censoring to subsequent therapy | through study completion, an average of 5 years
  Overall survival, AML-free survival and progressive-free survival censoring at subsequent therapy

OTHER OUTCOMES:
Patient reported outcomes | through study completion, an average of 5 years
  Patient reported outcomes according to the Myeloproliferative Neoplasm Safety Assessment Form Total Symptom Score which is a 10-item instrument designed to monitor clinically relevant symptoms among patients with myeloproliferative neoplasm. The score has possible range of 0 to 100.
Exploratory endpoints | through study completion, an average of 5 years
  Biomarkers including somatic mutations by targeted sequencing and BH3 profiling CD34+ cells and monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël ITZYKSON, MD/PhD, Principal Investigator — Hôpital Saint Louis; Pierre FENAUX, MD/PhD, Principal Investigator — Hôpital Saint Louis
Locations (24):
- France (24):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - Hôpital Avicenne, Bobigny
  - Hôpital privé Sévigné, Cesson-Sévigné
  - CHU de Grenoble, Grenoble
  - Hôpital Claude Huriez, Lille
  - CHRU de Limoges, Limoges
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - CHU de Montpellier - Hôpital Saint Eloi, Montpellier
  - CHU Hôtel Dieu, Nantes
  - Hôpital privé du Confluent SAS, Nantes
  - Hôpital Archet 1, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital Cochin, Paris
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre hospitalier Lyon sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Hôpital NOVO, Pontoise
  - Centre Hospitalier Annecy Genevois - Site d'Annecy, Pringy
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - IUCT oncopole, Toulouse
  - CHU de Tours - Hôpital Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No